CLINICAL TRIAL: NCT04833127
Title: Developing a Gender-Enhanced Pre-Exposure Prophylaxis (PrEP) Information-Motivational Workshop for Young South African Women
Brief Title: A Gender-Enhanced Pre-Exposure Prophylaxis (PrEP) Information-Motivational Workshop for Young South African Women
Acronym: Masibambane
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Medical Research Council, South Africa (Other); Brown University (Other)
Responsible Party: Principal Investigator, Susie Hoffman, Professor of Clinical Epidemiology (in Psychiatry), New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7682
Record Dates: First submitted 2021-03-21; First posted 2021-04-06 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: Pre-Exposure Prophylaxis, oral; South African; Adolescent girls and young women; HIV prevention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masibambane - Gender-Enhanced (Active Comparator): A virtual (online) group-based interactive Gender-Enhanced (GE) Workshop (using the WhatsApp® platform). The intervention has components that are conducted by participants on their own time as well as a "real-time" "live" interactive session.
  Interventions: Behavioral: Gender-Enhanced -- Masibambane
- Individually accessed (Other): In this condition women are given access to a PrEP video and to websites that provide information on PrEP and on contraception options.
  Interventions: Behavioral: Individually accessed

INTERVENTIONS:
Behavioral: Gender-Enhanced -- Masibambane — The intervention has components that provide PrEP information, provide information about HIV prevention and contraceptive options, prompt women to think about why they may be at risk for HIV, discuss women's sexual rights, and discuss how women can talk to their male partners about PrEP. The components are conducted by participants on their own time as well as during a "real-time" "live" interactive session with trained facilitators.
  Arms: Masibambane - Gender-Enhanced
Behavioral: Individually accessed — The intervention includes an individually-accessed online PrEP video and South African government websites on PrEP and on contraception options
  Arms: Individually accessed

SUMMARY:
This is a phase 1 pilot study to assess feasibility and acceptability and potential for impact of a gender-enhanced virtual group workshop focused on oral Pre-Exposure Prophylaxis (PrEP) as an HIV prevention method for young South African women. It was developed in collaboration with South African adolescent girls and young women (AGYW) aged 18-25. The investigators compared AGYW (N=100) assigned to the virtual group-based (GE) workshop to those assigned to an Individually Accessed (IA) condition in which women were given access to a PrEP video and to websites that provide information on PrEP and on contraception options. Investigators also evaluated the acceptability and feasibility of participant-driven recruitment (PDR). AGYW assigned to either intervention condition were invited to become Peer Health Advocates (PHAs), who were incentivized to talk to social network members and refer up to three to the intervention type the PHA attended. The aim was to assess if PDR is self-sustaining and is effective at reaching women who might not be reached in clinics.

DETAILED DESCRIPTION:
South African adolescent girls and young women (AGYW) remain at extraordinarily high risk of HIV infection. Oral pre-exposure prophylaxis (PrEP) has the potential to alter the epidemic in this vulnerable population, given that it is has been shown that if it is adhered to, oral PrEP can protect women from HIV infection. Yet, a critical question is whether AGYW will adopt and adhere to oral PrEP.

The investigators propose that two innovations can reach young, at-risk AGYW, inform them about PrEP and motivate them to use it: (1) introducing PrEP through a gender lens in a group workshop; and (2) participant-driven recruitment-recruiting women to attend the workshop by those who have already attended it. To inform intervention development, the investigators conducted six focus groups with sexually-active AGYW (aged 18-25), 8 qualitative interviews with focus group participants, and 20 qualitative interviews with men (10 HIV-positive, 10 HIV-negative or of unknown status) partnered with women in this age range that explored knowledge of, beliefs about, motivators for, and concerns about using PrEP in the context of gendered relationship dynamics and PrEP-related stigma. Guided by gender theory and the Information Motivation Behavior (IMB) model, and in collaboration with a Working Group of AGYW, a virtual (online) group-based Gender-Enhanced (GE) Workshop (using the WhatsApp® platform) was developed. The intervention has components that are conducted by participants on their own time as well as a "real-time" "live" interactive session and aims to provide PrEP information and address AGYW's barriers to using it. The goal of the intervention is to promote consideration of and uptake of PrEP.

In this phase 1 pilot study to assess feasibility and acceptability and potential for impact of the workshop, investigators compared AGYW (N=100) assigned to the virtual group-based (GE) workshop or to an Individually Accessed (IA) condition in which women were given access to a PrEP video and to websites that provide information on PrEP and on contraception options. To evaluate participant-driven recruitment (PDR), AGYW assigned to either condition were invited to become Peer Health Advocates (PHAs), who are incentivized to talk to social network members and refer up to three to the workshop type the PHA attended. Acceptability and feasibility of PDR were evaluated by assessing whether the method can be self-sustaining (i.e., on average >50% attendees become PHAs and >2 recruits/PHAs attend a workshop); and whether it reaches high-risk women and women who would not be captured by other methods of recruitment (percent who score high on HIV risk; percent who never tested or attended family planning). If promising, these approaches will be further tested in a larger study.

ELIGIBILITY:
Inclusion Criteria:

1. self-reported HIV-negative or unknown status
2. heterosexual vaginal or anal intercourse reported in the past 6 months
3. Is not currently taking PrEP or planning to begin PrEP
4. presently residing in eThekweni-metropolitan Durban
5. has private smart-phone access
6. Conversant in isiZulu or English
7. Willing to recruit other women (if in first group of participants);
8. (If recruited subsequent to first group): Recruited by a peer health advocate (someone the participant knew knew prior to being recruited)

Exclusion Criteria:

1. Overt signs of cognitive impairment
2. Was a participant in the previously conducted focus groups
3. If assigned to the online group intervention, unwilling to be audio-recorded

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 100 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- South African Medical Research Council, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrison A, Bhengu N, Miller L, Exner T, Tesfay N, Magutshwa S, Khumalo S, Bergam S, Hoffman S, Hanass-Hancock J. "You tell him that 'baby, I am protecting myself'": Women's agency and constraint around willingness to use pre-exposure prophylaxis in the Masibambane Study. Womens Health (Lond). 2022 Jan-Dec;18:17455057221087117. doi: 10.1177/17455057221087117. PMID 35306944
- [Background] Bergam S, Harrison AD, Benghu N, Khumalo S, Tesfay N, Exner T, Miller L, Dolezal C, Hanass-Hancock J, Hoffman S. Women's Perceptions of HIV- and Sexuality-Related Stigma in Relation to PrEP: Qualitative Findings from the Masibambane Study, Durban, South Africa. AIDS Behav. 2022 Sep;26(9):2881-2890. doi: 10.1007/s10461-022-03632-6. Epub 2022 Feb 26. PMID 35218452
- [Background] Fordjuoh J, Dolezal C, Bhengu N, Harrison AD, Exner TM, Hanass-Hancock J, Hoffman S. Peer-to-Peer Chain Recruitment for Enrolling Young South African Women into an HIV Pre-exposure Prophylaxis (PrEP) Intervention Study: How Did It Perform? AIDS Behav. 2024 May;28(5):1782-1794. doi: 10.1007/s10461-023-04256-0. Epub 2024 Feb 28. PMID 38416275
- [Background] Hanass-Hancock J, Bhengu N, Exner T, Magusthwa S, Harrison A, Dolezal C, Miller L, Bauman L, Hoffman S. Masibambane-Ladies Chat: Developing an Online Gender-Enhanced PrEP Information-Motivation Workshop for Young South African Women. AIDS Educ Prev. 2023 Feb;35(1):14-35. doi: 10.1521/aeap.2023.35.1.14. PMID 36735226
- See also: Publically-available website about the study — https://www.samrc.ac.za/intramural-research-units/gender-enhanced-prep-prep-project

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Met the goal
Units Other Than Participants: Recruitment seed
Period: Overall Study
Arm/Group | Masibambane - Gender-Enhanced | Individually Accessed
Started | 50; 8 Recruitment seed | 50; 8 Recruitment seed
Completed | 49; 8 Recruitment seed | 49; 8 Recruitment seed
Not Completed | 1; 0 Recruitment seed | 1; 0 Recruitment seed
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Masibambane - Gender-Enhanced | Individually Accessed | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 23 (2) | 22 (2) | 22 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Africa | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Have an Individual Counseling Session About PrEP.
Description: Percent of all participants who request and undergo an individual counseling session with the study nurse about the possibility of taking up PrEP. This behavioral measure will be documented by the study nurse
Time Frame: Immediate post-intervention up to 3 months after the intervention (i.e., as reported on the 3-month follow-up and nurse counselor log)
Measure: Count of Participants; unit: Participants
Arm/Group | Masibambane - Gender-Enhanced | Individually Accessed
Number analyzed (Participants) | 50 | 50
Participants | 28 | 28
Statistical Analysis 1: Comparison: Masibambane - Gender-Enhanced vs Individually Accessed; Test type: Equivalence — Null hypothesis: no difference between the groups; p = 1.0, GLM (logit link) with GEE — generalized linear models (GLM) and generalized estimating equations (GEE) for clustering within recruitment chain; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.56 to 1.80]
Statistical Analysis 2: Comparison: Masibambane - Gender-Enhanced vs Individually Accessed; Test type: Equivalence — Null H: No difference between the groups; p = 0.69, GLM (logit link) with GEE — GLM with GEE to account for clustering by recruitment chain; Adjusted for age, education, if has a main male partner, which differed between the two groups at baseline; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.62 to 2.07]

2. Secondary Outcome: Percent of Participants Who Undergo HIV-testing and Counseling (HCT).
Description: Percent of all participants who undergo HIV testing and counseling, using self-administered OraQuick, either on her own or with study nurse support. This behavioral measure will be documented by the study nurse.
Time Frame: Immediate post-intervention up to 3 months after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Masibambane - Gender-Enhanced | Individually Accessed
Number analyzed (Participants) | 50 | 50
Participants | 3 | 3
Statistical Analysis 1: Comparison: Masibambane - Gender-Enhanced vs Individually Accessed; Test type: Equivalence — Null hypothesis: No difference between the groups; p = 1.00, GLM with GEE; GLM with GEE accounting for clustering by recruitment chain; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.35 to 2.85]
Statistical Analysis 2: Comparison: Masibambane - Gender-Enhanced vs Individually Accessed; Test type: Equivalence — Null H: No difference between the 2 groups; p = 0.927, GLM (logit link) with GEE — GLM (logit link) with GEE to account for clustering by recruitment chain; adjusted for baseline differences in age, educational status, and whether has a primary male partner; Odds Ratio (OR) = .95, 95% CI 2-sided [0.31 to 2.90]

3. Secondary Outcome: Percent Taking up PrEP
Description: If participant is PrEP-eligible (HIV-negative) she initiates PrEP. This outcome will be based on self-report.
Time Frame: Immediate post-intervention up to 3 months after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Masibambane - Gender-Enhanced | Individually Accessed
Number analyzed (Participants) | 50 | 50
Participants | 8 | 5
Statistical Analysis 1: Comparison: Masibambane - Gender-Enhanced vs Individually Accessed; Test type: Equivalence — Null Hypothesis: No difference between the groups; p = 0.215, GLM (logit link) with GEE; Used GEE to account for clustering by recruitment chain; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.73 to 4.04]
Statistical Analysis 2: Comparison: Masibambane - Gender-Enhanced vs Individually Accessed; Test type: Equivalence — Null hypothesis: No difference between the groups; p = 0.295, GLM (logit link) with GEE; GEE used to account for clustering by recruitment chain; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.65 to 4.13] — adjusted for baseline differences in age, education, and whether has a main male partner

ADVERSE EVENTS:
Time Frame: up to the last assessment, at 3-months after the intervention.
Description: Adverse events in this study included:
  1. Violence or threat of violence to participant due to participating in HIV prevention activities
  2. Breach of confidentiality
  3. Stigmatization/discrimination due to participating in HIV prevention activities
  4. Serious emotional distress
Arm/Group | Masibambane - Gender-Enhanced | Individually Accessed
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Masibambane - Gender-Enhanced (N=50) | Individually Accessed (N=50)
violence from a partner (General disorders) | 1 | 0 — Participant reported an instance of intimate partner violence, not related to study participation

LIMITATIONS AND CAVEATS:
Pilot trial with sample size of 100 participants, designed to assess feasibility and acceptability rather than efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT04833127/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT04833127/SAP_001.pdf
  • Informed Consent Form (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT04833127/ICF_002.pdf